CLINICAL TRIAL: NCT05255224
Title: Predicting AF After Cardiac Surgery - the PARADISE Score. A Clinical Prediction Rule for Post-operative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Brief Title: PARADISE: Predicting AF After Cardiac Surgery
Acronym: PARADISE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: St. Bartholomew's Hospital (Other); University College, London (Other); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Brigham and Women's Hospital (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PID15669
Record Dates: First submitted 2022-02-07; First posted 2022-02-24 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation New Onset
Keywords: New Onset Atrial Fibrillation; Cardiac Surgery
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Patients admitted to Mass Brigham Hospitals for cardiac surgery from 1st January 1998 to 31st December 2020
  Interventions: Other: Not applicable as observational study
- Prospective: Patients admitted to Barts Health, Liverpool Heart and Chest Hospital, or Oxford University Hospitals NHS Foundation Trust for cardiac surgery between 1st October 2021 to 31st July 2023
  Interventions: Other: Not applicable as observational study

INTERVENTIONS:
Other: Not applicable as observational study — Not applicable as observational study

SUMMARY:
The PARADISE study aims to develop and validate prediction tools to identify patients at risk of Atrial Fibrillation (AF) after cardiac surgery.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is a common abnormal heart rhythm. AF causes the heart to beat irregularly and sometimes very rapidly. About 30-50% of patients develop AF after heart surgery. These patients stay longer on the Intensive Care Unit (ICU) after surgery, are more likely to develop complications and have a higher risk of dying. Avoiding AF is important.

Some drugs, including beta blockers and amiodarone may help prevent AF if given after surgery. However, these may also lead to complications (such as lung damage). It is therefore important to identify which patients are most likely to benefit from these treatments (i.e., where the benefits outweigh the risks). There are existing tools designed to predict the risk of suffering AF after heart surgery. However, they are unreliable and therefore not used in clinical practice. A modern, reliable risk prediction tool is needed.

The PARADISE study will develop and test new prediction tools to identify which patients are most at risk of developing AF after heart surgery. The investigators will focus our tools on those patients who most commonly develop AF, such as those who have had surgery to repair a valve or blood vessel in their heart.

To do this the investigators will:

* Review the medical literature and assemble a panel of medical experts to create a list of known factors that affect patients' risk of AF after heart surgery
* Use a large UK general practice database (CALIBER) to see whether the investigators can find new risk factors.
* Ask the expert panel to agree a list of known and new risks factors to be included in the prediction tool.
* Develop two new prediction tools using an existing American cardiac surgery database (the Partners research Database). The first will be used before surgery, the second immediately following surgery. Two models are needed as events during surgery may alter the risk of AF.
* Test how reliably our new tools predict which patients suffer AF after surgery, with data from large UK (United Kingdom) NHS (National Health Service) heart centres, one US Hospital (Brigham) and a UK clinical trial (Tight-K).
* The investigators will work with two charities (AF Alliance and StopAfib) to share our results with patients and the wider public.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or over
* Admitted to hospital for any cardiac surgery

Exclusion Criteria:

* Patients who have requested that their data not be used for research (e.g. NHS Opt-out)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 13684 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Model discrimination (c-statistic) to predict Atrial Fibrillation in external data set | Within 7 days of cardiac surgery
  Model discrimination (c-statistic) to predict Atrial Fibrillation in external data set
Model calibration (intercept) to predict Atrial Fibrillation in external data set | Within 7 days of cardiac surgery
  Model calibration (intercept) to predict Atrial Fibrillation in external data set
Model calibration (slope) to predict Atrial Fibrillation in external data set | Within 7 days of cardiac surgery
  Model calibration (slope) to predict Atrial Fibrillation in external data set

SECONDARY OUTCOMES:
Additional model performance metrics to predict Atrial Fibrillation in external data set | Within 7 days of cardiac surgery
  Model positive and negative predictive values, sensitivity and specificity to predict Atrial Fibrillation in external data set
Candidate risk factors for inclusion in new onset atrial fibrillation prognostic models | Within 7 days of cardiac surgery
  Candidate risk factors for inclusion in new onset atrial fibrillation prognostic models, identified through Systematic literature review and analysis of the CALIBER database using statistical and machine learning methods.
  For pre-operative model, the investigators will include patient information available up to the time of surgery. For the post-operative model, the investigators will also include patient information available up to 12 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Watkinson, MD, Principal Investigator — University of Oxford; Benjamin O'Brien, MD, Principal Investigator — Deutsches Herzzentrum der Charité
Locations (1):
- Critical Care Research Group, Nuffield Department of Clinical Neurosciences, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publicly available due to privacy and legal implications.

REFERENCES:
- [Derived] Bedford J, Fields KG, Collins GS, Lip GYH, Clifton DA, O'Brien B, Muehlschlegel JD, Watkinson PJ, Redfern OC. Atrial fibrillation after cardiac surgery: identifying candidate predictors through a Delphi process. BMJ Open. 2024 Sep 25;14(9):e086589. doi: 10.1136/bmjopen-2024-086589. PMID 39322590

DOCUMENTS (2):
  • Study Protocol (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT05255224/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT05255224/SAP_001.pdf